CLINICAL TRIAL: NCT00320736
Title: Effect of Nicotine Agonist Galantamine Added to High Potency Medications for Cognitive Function in Patients With Schizophrenia and Schizoaffective Disorder
Brief Title: Galantamine for Cognition in People With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Suffolk Mental Health Association (Other)
Collaborators: Janssen Medical Affairs (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORRC 20-01
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-05

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; cognitive function; cholinergic medication; nicotinic receptor agonist
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine

SUMMARY:
This study is a double-blind, placebo-controlled trial of the nicotinic receptor agonist, galantamine, for the improvement of memory and attention in people with schizophrenia and schizoaffective disorder. Twenty subjects on a stable dose of antipsychotic medications receive galantamine or identical placebo tablets for 8 weeks. Adverse events are screened for every week. Tests of memory, attention, and reward responsivity are performed at baseline and afer 8 weeks on medication. Clinical scales rating psychiatric symptoms are performed at the beginning, middle, and end of the trial.

DETAILED DESCRIPTION:
Background:

Galantamine is a novel acetylcholinesterase inhibitor that is also a positive allosteric modulator of nicotinic acetylcholine receptors. Galantamine has been shown to increase conductivity of nicotinic receptors through a binding site that is discreet from the acetylcholine receptor. There is minimal risk of overstimulation with positive allosteric modulators as they do not produce receptor depolarization but potentiate submaximal acetylcholine induced depolarization. Our hypothesis is that allosteric modulation of nicotinic acetylcholine receptors is a potentially important treatment strategy in schizophrenia. We propose a trial of galantamine augmentation of antipsychotic medication in the treatment of schizophrenia to test the following hypotheses.

Hypotheses:

1. Galantamine augmentation of antipsychotic treatment will be associated with improvement from baseline in performance on the cognitive battery: Stroop, Cornblatt CPT-IP, CDR Battery, letter number span, Grooved peg board, Tower of London, and Signal Detection Task.
2. Galantamine augmentation of high potency antipsychotic treatment will be well tolerated and associated with improvement from baseline in negative symptoms (SANS), depressive symptoms (CDSS) and impulsivity (PANSS aggression item).

Study Design:

Twenty adult subjects, aged 18-60, will be randomized, according to a double blind, parallel group design, to receive galantamine or identical placebo for 8 weeks. Subjects will begin with a dose of up to 8 mg twice per day for the first four weeks, then up to 16 mg twice per day for the next four weeks. Visits will be weekly to monitor medication compliance and medication side effects. Prior to beginning treatment, subjects will undergo a 1.5 hour training session to familiarize themselves with the CDR battery portion of the cognitive battery. Subjects will then be evaluated for symptoms of psychosis, depression, anxiety, smoking behavior and medication side effects with standard clinical rating scales that include the Schedule for Assessment of Negative Symptoms (SANS), Positive and Negative Symptom Scale (PANSS), Brief Psychiatric Rating Scale (BPRS), Calgary Depression Scale for Schizophrenia (CDSS), Abnormal Involuntary Movement Scale (AIMS), Simpson Angus Scale and Barnes Akathisia Scale, Fagerstrom Test of Nicotine Dependence, carbon monoxide measurement and smoking self report. Subjects who meet criteria for current depression or who have suicidal ideation will be excluded. Clinical rating scales will be performed at baseline and monthly. Tests of visual and spatial working memory, attention, motor skills, inhibition, and motivation will be performed at baseline and at 8 weeks. The cognitive battery will include tests of response inhibition (the 3-card Stroop), attention (Cornblatt continuous performance test identical pairs (CPT-IP) and CDR Battery), verbal memory (CDR Battery), working memory (letter-number span), non-verbal memory (CDR Battery), psychomotor ability (grooved peg board task), executive functioning (Tower of London), and motivation for reward (signal detection task). Blood will be drawn for antipsychotic levels, galantamine levels, and measurement of nicotinic receptor number at baseline and 8 weeks. Adverse events will be documented at each visit using an Adverse Events Tracking log. At baseline and week 8 carbon monoxide (CO) measurements will be used with self report to verify number of cigarettes smoked per day.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia or schizoaffective disorder depressed type with stable psychiatric symptoms, no active suicidal ideation
2. Age 18-60, inclusive
3. Stable medical conditions such as hypertension, non-insulin-dependent diabetes, hypothyroidism allowed
4. Treated with antipsychotic medications at a stable dose for > 4 weeks
5. Not treated with investigational medications in the past 30 days
6. Competent to provide informed consent
7. WRAT-3 IQ raw score greater than or equal to 35
8. Expired CO level < 9 ppm
9. Salivary cotinine level < 30 ng/ml
10. Non-smoker for at least 3 months

Exclusion Criteria:

1. Diagnosis of dementia, neurodegenerative disease or any other current Axis I DSM-IV diagnosis
2. Any unstable medical illness, asthma requiring daily treatment, severe COPD, active peptic ulcer disease, gastrointestinal bleeding, atrioventricular block, urinary outflow obstruction, history of epilepsy
3. Concurrent use of anticholinergic medications or use of cholinomimetic medications in the past month, such as cogentin, donepezil or clozapine
4. Alcohol or substance abuse in the past month (self-report and confirmed by chart)
5. Known allergy or hypersensitivity to galantamine
6. Current treatment with erythromycin or ketoconazole
7. Concurrent use of NSAIDs
8. Women of childbearing potential
9. History of suicide attempt in the past year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-01; Study Completion 2006-05

PRIMARY OUTCOMES:
Improvement from baseline in performance on the cognitive battery: Stroop, Cornblatt CPT-IP, CDR Battery, letter number span, Grooved peg board, Tower of London, and Signal Detection Task.

SECONDARY OUTCOMES:
Improvement from baseline in negative symptoms (SANS), depressive symptoms (CDSS) and impulsivity (PANSS aggression item).

CONTACTS AND LOCATIONS:
Overall Officials: A Eden Evins, MD, MPH, Principal Investigator — North Suffolk Mental Health Organization
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States